CLINICAL TRIAL: NCT04779593
Title: Impact of Transferrin Saturation Guided Maintenance Treatment on Quality of Life in HFE Haemochromatosis
Acronym: Quali-SAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35RC19_8985_Quali-SAT
Record Dates: First submitted 2021-02-02; First posted 2021-03-03 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Haemochromatosis
MeSH Terms: conditions — Hemochromatosis | interventions — Restraint, Physical; Biological Specimen Banks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients treated with bloodletting according to "transferrin saturation and serum ferritin".
  Interventions: Other: Clinical examination; Other: SF36 questionnaire; Other: AIMS2_SF questionnaire; Other: WOMAC questionnaire; Other: EQ-5D-5L questionnaire; Biological: Blood Sample Complete blood count; Biological: Blood Sample Iron panel; Biological: Blood Sample Fasting Glucose; Biological: Blood sample lipid panel; Biological: Blood sample liver panel; Biological: Blood sample C reactive protein; Biological: BioBank; Other: Medico-economical; Procedure: Bloodletting - experimental group
- control group (Active Comparator): Patients treated with bloodletting according to current guidelines "ferritin alone"
  Interventions: Other: Clinical examination; Other: SF36 questionnaire; Other: AIMS2_SF questionnaire; Other: WOMAC questionnaire; Other: EQ-5D-5L questionnaire; Biological: Blood Sample Complete blood count; Biological: Blood Sample Iron panel; Biological: Blood Sample Fasting Glucose; Biological: Blood sample lipid panel; Biological: Blood sample liver panel; Biological: Blood sample C reactive protein; Procedure: Bloodletting - control group; Biological: BioBank; Other: Medico-economical

INTERVENTIONS:
Other: Clinical examination — Clinical data will be recorded (general clinical examination, height, weight, blood pressure,heart beat, alcohol and tobacco consumption, antecedent) as well as concurrent medication at each follow-up visit.
Other: SF36 questionnaire — At D0, M12 and M24. This 36 item patient reported survey of patient's health is the most commonly used and validated health survey instrument for appraising quality of life.
  Items are grouped in 8 scaled scores exploring multiple dimension of global health (vitality, physical functioning, bodily pain, general health, perceptions, physical role functioning, emotional role functioning, social role functioning, mental health).
  Scoring will be performed as recommended by the SF-36 instruction manual to create the eight scale scores. Furthermore, these subscales sum to obtain the total SF-36 score and will be summarized into two composite scores (physical and mental quality of life).
Other: AIMS2_SF questionnaire — At D0, M12 and M24. The Arthritis Impact Measurement Scales 2 Short Form (AIMS2-SF) is a specific tool to measure changes in global health, pain, mobility and social function in patients with arthritis. It was described in 1992 in patients with rheumatoid arthritis and osteoarthritis and include 26 items that are summarized in scales according to a predefined scoring system: mobility, physical activity (walking, bending, lifting), dexterity, household activity (managing money and medications, housekeeping), social activities, activities of daily living, pain, depression, and anxiety. The French translation has been validated and this questionnaires has been widely used in the rheumatology field to assess quality of life of patients with arthritis. Because HFE related arthropathy is very similar to osteoarthritis this questionnaire is ought to be adequate in this setting.
Other: WOMAC questionnaire — At D0, M12 and M24. The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a widely used questionnaires specifically assessing lower limb (hips and knee) osteoarthritis. It measures five items for pain, two for stiffness and 17 for functional limitation and had been translated in French.
Other: EQ-5D-5L questionnaire — At D0, M12 and M24. The EQ-5D is a standardized instrument which evaluates the generic quality of life (http://www.euroqol.org/). It is a preference-based health-related quality of life measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The answers given to EQ-5D permit to find 243 health states that can be converted into utility score anchored at 0 for death and 1 for perfect health. EQ-5D is an instrument developed in Europe, widely used in cost-utility analysis. It has been validated in a representative sample of French population.
Biological: Blood Sample Complete blood count — Blood Sample Complete blood count at D0, M6, M12, M18 and M24/end follow-up visit
Biological: Blood Sample Iron panel — Blood Sample Iron panel (serum ferritin, serum iron and serum transferrin to determine transferrin saturation according to randomization group (at M6, M12 and M18) at D0, M6, M12, M18 and M24/end follow-up visit and at each bloodletting.
Biological: Blood Sample Fasting Glucose — Blood Sample Fasting Glucose at D0 and M24/end follow-up visit
Biological: Blood sample lipid panel — Blood sample lipid panel (total cholesterol, triglycerides, HDL, LDL) at D0 and M24/end follow-up visit
Biological: Blood sample liver panel — Blood sample liver panel (total bilirubin, Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Gamma-Glutamyl Transferase) at D0 and M24/end follow-up visit
Biological: Blood sample C reactive protein — Blood sample C reactive protein at D0 and M24/end follow-up visit
Procedure: Bloodletting - control group — Patients treated with bloodletting according to current guidelines (ferritin alone). Patient will undergo bloodletting with a goal of maintaining a serum ferritin equal or lower than 50 g/L according to current clinical practice guidelines (French and European).A first bloodletting will be performed at inclusion with the same volume as usually performed by the patients.Results of the biological test performed at this visit will guide the time schedule and volume of the next bloodletting according to randomization group. Time schedule and volume of bloodletting will be adjusted to biological results after each follow-up visit.
  Arms: control group
Biological: BioBank — Blood sample will be collected for BioBank at D0, M12 and M24.
Other: Medico-economical — Medico-economic data will be collected at each follow up visit.
Procedure: Bloodletting - experimental group — Patients treated with bloodletting according to "transferrin saturation and serum ferritin". Patients will undergo bloodletting with a goal of maintaining a serum transferrin saturation equal or lower than 50 % and a serum ferritin lower than the upper limit of the normal range (300 g/L for men and 200 g/L for women).A first bloodletting will be performed at inclusion with the same volume as usually performed by the patients.Results of the biological test performed at this visit will guide the time schedule and volume of the next bloodletting according to randomization group. Time schedule and volume of bloodletting will be adjusted to biological results after each follow-up visit.
  Arms: experimental group

SUMMARY:
Patients in maintenance treatment for HFE hemochromatosis since at least one year will be included in a two year study period and randomized in two groups experimental and control group. Because proton pump inhibitors are widely used as chronic medication, and because they can significantly modify iron absorption, patients will be stratified according to the use of proton pump inhibitors and gender. A first bloodletting will be performed at inclusion with the same volume as usually performed by the patients. Results of the biological test performed at this visit will guide the time schedule and volume of the next bloodletting according to randomization group (patients treated with bloodletting according to current guidelines "ferritin alone" versus patients treated with bloodletting according to "transferrin saturation and serum ferritin").Blood count and iron metabolism parameters will be performed at each bloodletting and follow-up visits. Time schedule and volume of bloodletting will be adjusted to biological results after each follow-up visit. Volume and schedule for bloodlettings will be determined according to guidelines specifically designed for this study to assure harmonization of treatment management, and centrally validated through the recording of the biological tests in the electronic Case Report Form which will provide the investigator with the volume and schedule of the next bloodletting. There will be two ways of treatment modification: either change of schedule or volume of bloodletting. Patients will undergo follow-up visit every six months with clinical examination, questionnaires at J0, M12 and M24 (SF-36; AIMS2-SF, WOMAC, EQ-5D-5L), and biological test. For health economics analysis, data will be obtained thanks to a dedicated extraction from SNDS database SNDS database will allow to gather hospital stays, visits, and other healthcare-related costs as well as vital status (date (month/year) of death) and cause of death. A de-identified copy of the clinical database, restricted to the relevant variables, will be sent for semideterministic matching purpose with SNDS extraction using four key variables: gender, same date (month/year) of birth, same date (day/month/year) of visit for bloodletting; pending, of course, regulatory authorization.

ELIGIBILITY:
Inclusion Criteria:

* - Patients treated with iron chelators;
* Patients treated with erythroid growth factors (erythropoietin);
* Patient with excessive alcohol consumption (> 20g/day and > 30 g/day for women and men respectively);
* Patients with chronic haematological condition;
* Patients having uncontrolled chronic blood loss (of digestive or gynaecological origin);
* Patients with chronic kidney failure;
* Patients with a diagnosis of cancer or history of cancer in the last year;
* Pregnancy or breast feeding.
* Patient who are included in another research protocol
* Adults legally protected (judicial protection, guardianship, or supervision), persons deprived of their freedom.
* with C282Y homozygous HFE hemochromatosis;
* having finished the initial phase of HFE hemochromatosis treatment and in maintenance treatment for at least one year;
* having signed an informed consent form.

Exclusion Criteria:

* Patients treated with iron chelators;
* Patients treated with erythroid growth factors (erythropoietin);
* Patient with excessive alcohol consumption (> 20g/day and > 30 g/day for women and men respectively);
* Patients with chronic haematological condition;
* Patients having uncontrolled chronic blood loss (of digestive or gynaecological origin);
* Patients with chronic kidney failure;
* Patients with a diagnosis of cancer or history of cancer in the last year;
* Pregnancy or breast feeding.
* Patient who are included in another research protocol
* Adults legally protected (judicial protection, guardianship, or supervision), persons deprived of their freedom.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The primary evaluation criteria is the Physical Component Score of the SF-36 questionnaire at the end of the study period (two years) | At Month 24
  The primary evaluation criteria is the Physical Component Score of the SF-36 questionnaire at the end of the study period (two years). Physical Component score of the SF-36 has been chosen because SF-36 it is a widely validated and reproducible questionnaire, and this component is best susceptible to reflect both fatigue and joint involvement.

SECONDARY OUTCOMES:
the AIMS2- SF (short form of the Arthritis Impact Measurement Scales 2) questionnaire | at Day 0, Month 12 and Month 24 follow-up visit
  Assessment of Arthropathy and joint pain related quality of life as assessed by the AIMS2- SF (short form of the Arthritis Impact Measurement Scales 2) questionnaire throughout the study, as performed at J0, M12 and M24 follow-up visit (every 12 months).
the WOMAC (Western Ontario and McMaster Universities Arthritis Index) questionnaire | at Day 0, Month 12 and Month 24 follow-up visit
  Assessment of Arthropathy and joint pain related quality of life as assessed by the WOMAC (Western Ontario and McMaster Universities Arthritis Index) questionnaire throughout the study, as performed at J0, M12 and M24 follow-up visit (every 12 months).
Evolution of the Mental Component Score of the SF-36 questionnaire | At Month 24
  Evolution of the Mental Component Score of the SF-36 questionnaire between inclusion and the end of the study period (two years).
Evolution of the Physical Component Score of the SF-36 | at Day 0, Month 12 and Month 24 follow-up visit
  Evolution of the Physical Component Score of the SF-36 throughout the study, as performed at J0, M12 and M24 follow-up visit (every 12 months).
Evolution of the Mental Component Score of the SF-36 | at Day 0, Month 12 and Month 24 follow-up visit
  Evolution of the Mental Component Score of the SF-36 throughout the study, as performed at J0, M12 and M24 follow-up visit (every 12 months).
Evolution of of the EQ-5D-5L score | at Day 0, Month 12 and Month 24 follow-up visit
  Evolution of of the EQ-5D-5L score throughout the study, as performed at J0, M12 and M24 follow-up visit (every 12 months).
Evolution of Serum ferritin and serum transferrin saturation | Day 0, Month 6, Month 12, Month 18 and Month 24/follow-up visit
  Evolution of Serum ferritin and serum transferrin saturation determined at each follow-up visit (every 6 months).
Occurrence of anaemia | Day 0, Month 6, Month 12, Month 18 and Month 24/follow-up visit
  Occurrence of anaemia defined as haemoglobin lower than 11g/dL at any follow-up visit.
Occurrence of malaise | At Month 24
  Occurrence of malaise after a bloodletting procedure
Total number of phlebotomy performed | At Month 24
  Total number of phlebotomy performed by each patient during the study period.
Incremental Cost-Effectiveness Ratio | At Month 24
  Incremental Cost-Effectiveness Ratio (ICER) defined as the cost for QALY gained in the "transferrin saturation + ferritin" strategy versus "ferritin alone" strategy.

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Hopital Avicenne, Bobigny
  - CHU Dupuytren, Limoges
  - GHBS site du Scorff, Lorient
  - GHRMSA - Hôpital Emile Muller, Mulhouse
  - CHR Orléans, Orléans
  - Hôpital Européen Georges Pompidou, Paris
  - CHU Rennes, Rennes
  - CH Yves le Foll, Saint-Brieuc
  - CH de St Malo, St-Malo
  - Hôpital Rangueil, Toulouse
  - Centre hospitalier Bretagne Atlantique, Vannes
  - Hôpital Paul Brousse, Villejuif